CLINICAL TRIAL: NCT06409403
Title: Study on Clinical Application of Robotic Technique
Brief Title: Study on Effect of Robotic Versus Laparoscopic Surgical Technology on Genitourinary Function After Total Mesorectal Excision for Rectal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: general surgery 3 (Other)
Responsible Party: Sponsor-Investigator, general surgery 3, Director of Gastrointestinal Surgery, The Third Xiangya Hospital of Central South University
Organization: The Third Xiangya Hospital of Central South University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YB2017
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- da Vinci robotic TME (Experimental)
  Interventions: Device: clinical application of robotic technique
- Microhands robotic TME (Experimental)
  Interventions: Device: clinical application of robotic technique
- laparoscopic surgery TME (Active Comparator)
  Interventions: Device: clinical application of robotic technique

INTERVENTIONS:
Device: clinical application of robotic technique — effect of various surgical technique on clinical efficacy of TME

SUMMARY:
Intraoperative pelvic autonomic nerve (PAN) injury is the dominant reason for genitourinary malfunction after total mesorectal excision (TME), particularly in low rectal tumours. TME necessitates meticulous, sharp dissection with an awareness of the PAN pathway. In particular, laparoscopic TME (L-TME) is technically difficult and requires advanced laparoscopic surgical skills. Comparing with the conventional laparoscopic approach, 3D vision, surgeon-manipulated camera systems, and multi-degree-of-freedom robotic instruments facilitate identification and preservation of the PAN during robotic-assisted TME (R-TME), theoretically facilitating favourable recovery of postoperative genitourinary function. Previous studies have mostly focused on the impact of advanced robotic technologies on postoperative functions. However, in addition to robotic surgical technology, postoperative function is impacted by multiple other intricate factors, such as oncology, comorbidities, postoperative complications, and adjuvant chemoradiotherapy. Consequently, the superiority of robotic surgery in terms of recovery of postoperative genitourinary function has been controversial in previous studies. Hence, to comprehensively evaluate the effect of robotic technology on postoperative genitourinary function, we conducted a prospective controlled study comparing the conventional approach and robotic surgery.

ELIGIBILITY:
Inclusion Criteria: (i) lesions that were determined by histopathological examination and were staged preoperatively using pelvic MRI and CT scans; (ii) patients aged ≥18 and ≤ 75 years; and (iii) American Society of Anesthesiology (ASA) class ≤3

Exclusion Criteria: Benign prostate hyperplasia, previous bladder or prostate surgery, severe sexual dysfunction (International Index of Erectile Function (IIEF) score <10 or Female Sexual Function Index (FSFI) score ≤26.55), urgent operation, simultaneous or heterochronous multiple primary rectal tumours, distant metastasis, or other severe cardiopulmonary complications.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
International Prostate Symptom Score (IPSS) | preoperation，1、3、6、12 months after operation
  evaluation of genitourinary function

SECONDARY OUTCOMES:
International Index of Erectile Function (IIEF) | preoperation，1、3、6、12 months after operation
  evaluation of genitourinary function
Female Sexual Function Index (FSFI) | preoperation，1、3、6、12 months after operation
  evaluation of genitourinary function
operative time | perioperative
  operative outcomes
blood loose | perioperative
  operative outcomes
conversion | perioperative
  operative outcomes
retrieved lymph nodes | perioperative
  operative outcomes
complete TME specimens | perioperative
  operative outcomes
circumferential resection margins (CRMs) | perioperative
  operative outcomes
complication | perioperative
  operative outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No